CLINICAL TRIAL: NCT05305976
Title: Remote Physiotherapy Application to Protect Physical Health in Duchenne Muscular Dystrophy
Brief Title: Telerehabilitation in Duchenne Muscular Dystrophy
Acronym: Duchenne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Arzu ERDEN, Associate Professor, Karadeniz Technical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KTU_FTR_AE_01
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; telerehabilitation; satisfaction
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Personal Satisfaction | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Grup 1: Ambulant Group Grup 2: Non-ambulant Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambulant Group (Experimental): Individuals unable to walk according to the Brooke Function Classification System
  Interventions: Other: Telerehabilitation
- Non-ambulant Group (Experimental): Individuals who can walk according to the Brooke Function Classification System
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — The 8 week exercise program with telerehabilitation

SUMMARY:
Duchenne Muscular Dystrophy (DMD) is a progressive inherited disease that affects the muscles and causes functional limitations to varying degrees. It is vital to start physiotherapy follow-ups immediately after diagnosis. Patients with DMD are among the most vulnerable groups who have problems in accessing physiotherapy services during the COVID-19 pandemic. The aim of the study was to investigate the effects of the telerehabilitation program developed to protect the physical health of patients with DMD and not to interrupt their follow-up.

DETAILED DESCRIPTION:
Forty two patients with DMD were included in the study. 30 of them were ambulant in group 1, and 12 were non-ambulant in group 2. Physiotherapy assessments were performed blindly before the program started. According to the functional levels of the individuals, 2 groups were formed. 9 physiotherapists applied the tele-rehabilitation program for 24 session (3 days in a week).

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate verbally and visually
* Older than 5 years old

Exclusion Criteria:

* The children who had undergone any surgical operations in the past 6 months,
* Having a severe cognitive and breathing impairment
* Using mechanical ventilator continually or intermittent
* Having a febrile infection

Min Age: 5 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Functional level | Before the intervention, up to one month
  Brooke Function Classification System
Socio-demographics | Before the intervention, up to one month
  gender, body weight, height
Walking test (Before intervention) | Before the intervention, up to one month.
  The distance of 10 m was determined in a suitable indoor environment.
Walking test (After intervention) | After the intervention, average two weeks.
  The distance of 10 m was determined in a suitable indoor environment.
Time to stand up from the supine position (Before intervention) | Before the intervention, up to one month.
  The time to stand up from the supine position was recorded.
Time to stand up from the supine position (After intervention) | After the intervention, average two weeks.
  The time to stand up from the supine position was recorded.
Modified upper extremity performance test (Before intervention) | Before the intervention, up to one month.
  Flexion the shoulder to 90 degrees, flexion the shoulder above 90 degrees (above eye level), abduction of the shoulder 90 degrees, abduction of the shoulder above 90 degrees, doing the same movements with weight, bringing the empty glass to the mouth in a sitting position, bringing the full glass to the mouth
Modified upper extremity performance test (After intervention) | After the intervention, average two weeks.
  Flexion the shoulder to 90 degrees, flexion the shoulder above 90 degrees (above eye level), abduction of the shoulder 90 degrees, abduction of the shoulder above 90 degrees, doing the same movements with weight, bringing the empty glass to the mouth in a sitting position, bringing the full glass to the mouth
Endurance (Before intervention) | Before the intervention, up to one month.
  The number of knee extensions and elbow flexions they can do in sitting position in 30 seconds
Endurance (After intervention) | After the intervention, average two weeks.
  The number of knee extensions and elbow flexions they can do in sitting position in 30 seconds
Pulmonary Dysfunction Test (Before intervention) | Before the intervention, up to one month.
  Value when the patient counts audibly in a single expiration after maximum inspiratory effort
Pulmonary Dysfunction Test (After intervention) | After the intervention, average two weeks.
  Value when the patient counts audibly in a single expiration after maximum inspiratory effort

SECONDARY OUTCOMES:
Patient Satisfaction Survey | After the intervention average two weeks
  General satisfaction, internet/connection, physiotherapist's guidance, timing, level of knowledge, reassurance, comfort, knowledge/advice, level of satisfaction with information clarity

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Ortahisar, Turkey (Türkiye)